CLINICAL TRIAL: NCT03997318
Title: JPN1: A Confirmatory, Bridging, Double-Blind, Randomized, Controlled Trial in Japan Comparing the Safety and Efficacy of AMDC-USR With Placebo in Female Subjects With Stress Urinary Incontinence
Brief Title: Japanese Bridging Study of Autologous Muscle Derived Cells Compared to Placebo for Female Urinary Sphincter Repair(JPN1)
Acronym: JPN1
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study not initiated due to business decision, no participants enrolled.
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-09
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence; Urinary Stress Incontinence; Lower Urinary Tract Symptoms; Urinary Bladder; Urinary Tract Diseases; Bladder; Urinary Leak; Urine Leak; Bladder Leak; Urethra; Urethral Spincter
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Lower Urinary Tract Symptoms; Urologic Diseases; Nocturnal Enuresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AMDC-USR (Experimental): AMDC-USR is the study product (Autologous Muscle Derived Cells for Urinary Sphincter Repair).
  Interventions: Biological: AMDC-USR
- Placebo (Placebo Comparator): Placebo control is the vehicle solution used for the study product.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AMDC-USR — Autologous Muscle Derived Cells for Urinary Sphincter Repair
  Arms: AMDC-USR
Other: Placebo — Placebo control is the vehicle solution used for the study product.
  Arms: Placebo

SUMMARY:
This is a confirmatory/bridging study to evaluate the efficacy and safety of Autologous Muscle Derived Cells for Urinary Sphincter Repair (AMDC-USR) compared with placebo in the treatment of stress urinary incontinence (SUI) in adult Japanese female subjects. Half of the participants will receive AMDC-USR (injections with cells) and the other half will receive placebo.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is the accidental loss of urine due to physical activity, such as laughing, coughing, or sneezing. Autologous Muscle Derived Cells for Urinary Sphincter Repair (AMDC-USR) involves a medical procedure in which a participant's own muscle cells are collected, processed, and then injected into the tissues of the urinary passage.

This is a double-blind randomized study, which means neither the participant, nor the study doctor will know which treatment group the participant will be in. Participants who are randomly chosen to receive injection with placebo will have the option to receive an injection with their cells after completion of the blinded portion of their study participation (12 months).

This trial was designed as a confirmatory Phase III study to bridge efficacy and safety data from the Japanese population to the current Phase III global trial for AMDC-USR (CELLBRATE, NCT03104517).

ELIGIBILITY:
Inclusion Criteria:

* Adult female patient 50 to 75 years of age who has primary and moderate-to-severe symptoms of SUI for at least 6 months, as confirmed by patient medical history and clinical symptoms, including a focused incontinence evaluation.
* Must be willing and able to comply with the study procedures, be mentally competent and able to understand all study requirements, and must agree to read and sign the informed consent form prior to any study-related procedures.
* Must have completed 100% of the screening 3-day diary evening reports.

Exclusion Criteria:

* Patient has symptoms of only urge incontinence as confirmed by basic evaluation of etiology from a patient medical history, including a focused incontinence history.
* Patient has symptoms of mixed urinary incontinence where urge incontinence is the predominant factor.
* Patient has had stress urinary incontinence symptoms less than 6 months prior to signing the informed consent.
* Patient has not previously attempted conservative treatment prior to signing the informed consent. (Examples of conservative treatment include behavior modifications, bladder exercises, biofeedback, pelvic floor muscle therapy, etc.)
* Patient BMI ≥ 35.
* Patient routinely has more than 2 episodes of awakening to void during normal sleeping hours.
* If taking a medication known to affect lower urinary tract function, including but not limited to, anticholinergics, beta 3 adrenergic receptor agonists, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitor (SNRI) or selective serotonin reuptake inhibitor (SSRI) antidepressants, diuretics, or alpha-adrenergic blockers, patient cannot be maintained on a stable dose and/or frequency of medication (including diuretics), cannot be maintained on a stable dose and/or frequency for at least 2 weeks prior to screening or is likely to change during the course of the study.
* History of cancer in pelvic organs, ureters, or kidneys.
* Patient is pregnant, lactating, or plans to become pregnant during the course of the study.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of leaks due to stress incontinence episodes, as recorded in a diary. | 12 months
  Stress leak frequency

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kaufman, M.D., Ph.D., Principal Investigator — Vanderbilt University Medical Center, Department of Urologic Surgery

IPD SHARING:
Plan to Share IPD: No